CLINICAL TRIAL: NCT04500184
Title: Can Exercise-based Cardiac Rehabilitation Increase Physical Activity in Patients Who Undergoing Totally Thoracoscopic Ablation?
Brief Title: Exercise-based Cardiac Rehabilitation After Thoracoscopic Ablation in Patients With Persisent Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Dong Seop Jeong, Clinical professor, Samsung Medical Center
Other Study IDs: samsungmc_rehab_TTA
Record Dates: First submitted 2020-07-24; First posted 2020-08-05 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-07

CONDITIONS: Atrial Fibrillation, Persistent; Cardiac Rehabilitation; Cardiopulmonary Fitness
MeSH Terms: conditions — Atrial Fibrillation | interventions — Cardiac Rehabilitation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exercise group: patients who underwent cardiac rehabilitation
  Interventions: Other: cardiac rehabilitation
- Control group: patients who did not undergo cardiac rehabilitation

INTERVENTIONS:
Other: cardiac rehabilitation — rehabilitation performed by professional trainers
  Groups: Exercise group

SUMMARY:
Thoracoscopic ablation is a promising treatment of persistent atrial fibrillation. However, the postoperative rehabilitation is very important to prevent early recurrence of atrial arrhythmia. The purpose of this study is to evaluate the efficacy of professional cardiac rehabilitation in patients after thoracoscopic ablation.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent thoracoscopic ablation due to persisent atrial fibrillation

Exclusion Criteria:

* below 18 years
* over 80 years old
* malignancy
* pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent thoracoscopic ablation were included. cardiac rehabilitation was performed according to the willingness of each patients.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Recurrence of atrial fibrillation | every 6 months for 1 year
  Atrial fibrillation recurrence after surgical treatment
functional recovery | 6 months after intervention
  exercise capacity and international physical activity questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Dong Seop Jeong, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea